CLINICAL TRIAL: NCT00127361
Title: Evaluation of Continuous Support in Labor
Brief Title: Study of Having a Female Friend as Labor Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Peters University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAC-1998
Record Dates: First submitted 2005-08-04; First posted 2005-08-05 (Estimated); Last update posted 2005-08-23 (Estimated); Status verified 2005-04

CONDITIONS: Pregnancy; Delivery, Obstetric
Keywords: doula; caregivers; labor support; being with woman; continuous labor support; maternal outcomes; Parturition

INTERVENTIONS:
Behavioral: doula training

SUMMARY:
The purpose of this study was to compare labor outcomes in women accompanied by an additional support person (doula group) with outcomes in women who did not have this additional support person (control group).

The current study was designed with the benefits of continuous labor support in mind as well as the need for a cost-effective, affordable program to provide those services for low-income women. Its purpose was to evaluate the effects of continuous labor support provided by a female companion of the pregnant person's choosing who, with the mother, had participated in an educational program to teach her how to provide continuous labor support.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the influence of a female companion in labor who had been chosen by a nulliparous, underinsured, low-income woman and who had received brief training in supportive labor techniques. The objective was to compare labor outcomes, specifically cesarean section rates, in women accompanied by this additional support person (doula group) with outcomes in women who did not have this additional support person (control group).

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous (never given birth before)
* Singleton pregnancy
* Vertex presentation
* Low risk pregnancy
* Has a female friend willing to be a doula

Exclusion Criteria:

* Placenta previa
* Abruptio placenta
* Multiple pregnancy
* Breech presentation
* Planned operative delivery

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 600
Dates: Start 1998-01; Study Completion 2003-02

PRIMARY OUTCOMES:
Length of labor
type of delivery
type and timing of analgesia/anesthesia

SECONDARY OUTCOMES:
Birthweight
neonatal Apgar score at 1 and 5 minutes after birth

CONTACTS AND LOCATIONS:
Overall Officials: Della A Campbell, PhDc, Principal Investigator — Saint Peters University Hospital
Locations (1):
- Saint Peters University Hospital, New Brunswick, New Jersey, United States